CLINICAL TRIAL: NCT00391937
Title: Efficacy of a New Resurfacing Hip Prosthesis. A Multicenter, Prospective, Randomized, Controlled Study
Brief Title: Efficacy of a New Resurfacing Hip Prosthesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, maaike vissers, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-DP-001
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Osteoarthritis, Hip
Keywords: "resurfacing hip" [MESH]; "conventional position method"; "surgery, computer-assisted" [MESH]
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Hip Prosthesis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): ASR prosthesis placed using CAS
  Interventions: Device: Articular Surface Replacement (ASR) hip prosthesis
- 2 (Active Comparator): ASR prosthesis placed by conventional method
  Interventions: Device: Articular Surface Replacement (ASR) hip prosthesis

INTERVENTIONS:
Device: Articular Surface Replacement (ASR) hip prosthesis — a DePuy ASR™ primary resurfacing femoral and acetabular component (DePuy International Ltd, Leeds, UK). The cement that will be used is one dose of DePuy SmartSet® GHV 40 gram, a high-viscosity cement with gentamycin (DePuy CMW, Blackpool, UK). Instrumentation includes standard ASR™ instruments and Ci™ Software for DePuy ASR™ System1.0.

SUMMARY:
The purpose of this study is to compare the articular surface replacement (ASR) prosthesis placed by the conventional positioning method and the ASR prosthesis placed by 'computer assisted surgery' (CAS) in variation between pre planned position of the femoral component and the actual position of the femoral component of the prosthesis. The hypothesis is that this variation is larger with the conventional positioning method than when CAS is used.

DETAILED DESCRIPTION:
For patients who suffer from end stage of osteoarthritis of the hip, a joint replacement could result in an obvious improvement of the quality of life. However, because of the life expectation and high level of activity of young and active patients, the conventional total hip replacement does not offer an optimal solution.

An alternative to a total hip replacement in young and active patients is the resurfacing hip prostheses. The articular surface replacement (ASR) hip prostheses can be placed by the conventional positioning method and by using 'computer assisted surgery' (CAS). The hypothesis is that the positioning of the femoral component by the conventional positioning method will show a larger variation between pre planned and actual position than when CAS is used.

This study will compare the results of those who had an ASR prosthesis placed by the conventional positioning method with those patients in whom the ASR prosthesis was placed using CAS.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≤ 60 years, and women aged ≤ 55 years
* Presence of evident clinical and radiological osteoarthritis of the hip, indicated for a joint replacement surgery

Exclusion Criteria:

* Evident osteoporosis
* Active local or systemic infection
* Clinical manifestation of vascular deficiency of the lower extremity
* Pathological condition of the acetabulum
* Presence of evident clinical and radiological avascular necrosis of the femoral head, hip dysplasia, slipped capital femoral epiphysis, Legg-Calve- Perthes disease
* Rheumatoid arthritis
* Extreme varus position (neck-shaft angle < 110º)
* Presence of femoral cyst > 1 cm in diameter
* Previous hip surgery
* Presence of bilateral hip pathology, which may lead to joint replacement surgery within 1 year
* Presence of a THR at the contra lateral site less than 6 months post- operatively or patients with a THR at the contra lateral site with a poor function of the hip
* BMI> 30 kg/m2
* Renal deficiency (creatine > 115 μmol/l for men and > 90 μmol/l for women)
* Medically proven metal allergy
* Request of patient to correct an existing leg length discrepancy
* Head-neck ratio < 1
* Use of steroids, and/or immunosuppressive medication
* Alcoholism
* Patients from which it is not sure that they will be able to attend the follow-up measurements
* Insufficient command of the Dutch language, spoken and/of written

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2006-10; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
pre planned position of the femoral component preoperatively (stem-shaft-angle) | within 8 weeks before surgery
actual position of the femoral component postoperatively (stem-shaft-angle) | within one week after surgery

SECONDARY OUTCOMES:
Harris Hip Score | preoperatively and at 6 weeks, 3, 12, 24 and 36 months postoperatively
Hip pain | preoperatively and at 6 weeks, 3, 12, 24 and 36 months postoperatively
Assessments of the position of femoral component (biomechanical parameters) at the X-rays | preoperatively, during the clinical phase and at 6 weeks, 3, 12, 24 and 36 months postoperatively
Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) | preoperatively and at 6 weeks, 3, 12, 24 and 36 months postoperatively
Percentage of dynamic and static activities measured by the Rotterdam Activity Monitor (RAM) | preoperatively and at 3 and 6 months postoperatively
Quality of life | preoperatively and at 6 weeks, 3, 12, 24 and 36 months postoperatively
Early complications | within 3 months after surgery
Later complications | longer than 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: JAN Verhaar, PhD MD, Study Director — Erasmus Medical Center
Locations (6):
- Netherlands (6):
  - Laurentius Hospital, Roermond, Limburg
  - Maxima Medical Center, location Eindhoven, Eindhoven, North Brabant
  - Medical Center Haaglanden, location Antoniushove, Leidschendam, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Medical Center Haaglanden, location Westeinde Hospital, The Hague, South Holland
  - Oosterschelde Hospital, Goes, Zeeland

REFERENCES:
- [Derived] Koper MC, Reijman M, van Es EM, Waarsing JH, Koot HWJ, Keizer SB, Jansen I, van Biezen FC, Verhaar JAN, Bos PK. No added value for Computer-Assisted surgery to improve femoral component positioning and Patient Reported Outcomes in Hip Resurfacing Arthroplasty; a multi-center randomized controlled trial. BMC Musculoskelet Disord. 2019 Oct 25;20(1):473. doi: 10.1186/s12891-019-2883-7. PMID 31651318